CLINICAL TRIAL: NCT00521391
Title: Physical Activity as an Aid for Smoking Cessation: a Randomized Controlled Trial
Brief Title: Physical Activity as an Aid for Smoking Cessation
Acronym: PHASMO
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: End of the recruitment
Sponsor: University of Lausanne Hospitals (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3200-0637200; 3200-0637200
Record Dates: First submitted 2007-08-24; First posted 2007-08-27 (Estimated); Last update posted 2007-08-27 (Estimated); Status verified 2007-08

CONDITIONS: Tobacco Dependence; Cardiovascular Diseases; Physical Activity
Keywords: smoking cessation; nicotine; physical activity
MeSH Terms: conditions — Tobacco Use Disorder; Cardiovascular Diseases; Motor Activity; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): a tailored physical activity intervention involving moderate-intensity exercise
  Interventions: Other: Allez Hop
- B (No Intervention)

INTERVENTIONS:
Other: Allez Hop — a tailored physical activity intervention involving moderate-intensity exercise
  Arms: A

SUMMARY:
Including a tailored moderate-intensity physical activity intervention in a standard smoking cessation treatment program (pharmaceutical treatment and counseling) increases the chances of quitting and reduces nicotine withdrawal symptoms, negative moods, stress, and weight gain.

DETAILED DESCRIPTION:
The main objective is to determine whether a tailored physical activity intervention involving moderate-intensity exercise is an added value to a standard smoking cessation intervention in term of likelihood of smoking abstinence.

The secondary objectives are 1) to determine whether this tailored physical activity intervention prevents weight gain, reduces withdrawal symptoms, stress and improve mood and self-confidence in quitting; 2) to assess the effect of this tailored physical activity intervention on body composition and leptin concentration.

We assess this intervention in a randomized controlled trial of 600 sedentary adults regular smokers recruited from the community allocated into one of the two groups (intervention group vs. control group) during a 10-week period and 3 follow-up visits (6 and 12 months follow-up). All subjects (intervention and control groups) participate in a smoking cessation program composed of a pharmacological treatment (including nicotine replacement therapy) and counseling. The intervention group attend the 10-week physical activity program blending moderate-intensity exercise (Swiss nationwide implemented program entitled "Allez Hop!") and lifestyle physical activity and the control group a 10-week health education program to ensure equal contact condition.

ELIGIBILITY:
Inclusion Criteria:

1. Current daily smoker >10 or more cigarettes per day
2. Having smoked (on average > 10 cigarettes/day) regularly for at least 3 years
3. Age between 18 and 65 years
4. Sedentary lifestyle defined as less than 20 minutes a day of moderate-intensity physical assessed by the Swiss Baseline Questionnaire.

Exclusion Criteria:

1. Current pharmacological agent use to quit smoking
2. Medical problems that would alter training responses: arthritis, heart disease, and orthopedic problems
3. Presence of an unstable medical condition
4. Current or recent major cardiovascular event, such as recent myocardial infarction (>12 months) or stroke, angina pectoris, major arrhythmia
5. Current psychiatric illness
6. Alcohol (> 4 drinks/day for men and > 3 drink/d. for women), or/and other substance abuse
7. Current or planned pregnancy
8. Systematic skin disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2003-04; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
smoking cessation | 12 months

SECONDARY OUTCOMES:
weight change | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Cornuz, MD, Principal Investigator — University of Lausanne

REFERENCES:
- [Derived] Gonseth S, Locatelli I, Bize R, Nussle S, Clair C, Pralong F, Cornuz J. Leptin and smoking cessation: secondary analyses of a randomized controlled trial assessing physical activity as an aid for smoking cessation. BMC Public Health. 2014 Sep 3;14:911. doi: 10.1186/1471-2458-14-911. PMID 25187423
- [Derived] Bize R, Willi C, Chiolero A, Stoianov R, Payot S, Locatelli I, Cornuz J. Participation in a population-based physical activity programme as an aid for smoking cessation: a randomised trial. Tob Control. 2010 Dec;19(6):488-94. doi: 10.1136/tc.2009.030288. Epub 2010 Aug 25. PMID 20798023